CLINICAL TRIAL: NCT07058701
Title: Serum Instant Anti-Redness Efficacy Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: C24005025
Record Dates: First submitted 2025-06-18; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Female; Redness
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Serum (Other)
  Interventions: Other: Investigational Serum, Standard Cleanser; Device: Infrared Light for Redness Induction on Face
- Group Blank (Other)
  Interventions: Device: Infrared Light for Redness Induction on Face

INTERVENTIONS:
Other: Investigational Serum, Standard Cleanser — Mode of Group Serum application : On-site single use
  Standard cleanser + Investigational Serum (random half-face) [FLA #2039128 50]
  - subjects should wash face with standard cleanser [FLA #730457 36] on site before measurements.
  The technician will apply the Investigational Serum [FLA #2039128 50] on the subject's half face (according to the Annex 11.6) at the test site, keep another half face as blank control.
  Arms: Group Serum
Device: Infrared Light for Redness Induction on Face — Infrared light has high radiation frequency, its permeability is strong, the wavelength of infrared light can penetrate the human dermis to promote blood circulation and induce skin redness.The redness induction process will be done after baseline measurements for each subject.The subject's face was exposed at a distance of 20cm from infrared lamp for minimum 5 - 10 minutes at a temperature of 30-40°C and a wavelength of 760-5000 nm. In general, the skin will not be burned during the induction process. Due to individual differences, if the subjects cannot tolerate or feel uncomfortable during the process, the investigators will stop the process according to the situation; If there is any burn during the process, the on-site dermatologist will treat it in time, and the subject needs to follow the dermatologist's advice for follow-up treatment.
  Infrared light type: PHILIPS, IR250 RH IR2, 230-250V, 250W, wave length 760-5000nm, T 30~40°C

SUMMARY:
This study is a mono-centric, om-site use, random half-face application, blank control study. 64 female adult subjects will be enrolled and divided into 2 groups in the study, recruited according to inclusion and non-inclusion criteria listed above. At least 30 subjects for each group should complete the test in this 1 visit study.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women aged from 20-40 years old.
2. Self-declared mild sensitive skin.
3. Regular users of cleanser, Serum, moisturizer and sunscreen product.
4. Self-declare with skin concerns of redness and easy to flushing.
5. Willing to be exposed to infrared light on the facial skin to induce facial redness (can tolerate heat sensation on the face).
6. Clinical grading of skin redness(visual) ≥ 4 after infrared light[2] induction (5-10 mins) by dermatologist.
7. No disagreement of dermatologist because of other reasons that exclude the participation of the subject.
8. In general good health at the time of the study.
9. Willing and able to participate as evidenced by signing of informed consent and photo release form.
10. Must be willing to comply with all study protocol requirements (pay attention to: only use the provided product during the study, not take topical or oral treatment like retinol, hormone, anti-oxidant health-care products which may impact the efficacy of study).

Exclusion Criteria:

1. Allergic to infrared light
2. Pregnant or breast-feeding woman or woman planning pregnancy during the study.
3. Subject deprived of rights by a court or administrative order.
4. Major subject to a guardianship order.
5. Subject residing in a health or social care establishment.
6. Patient in an emergency setting.
7. Subject with a skin disease in the test areas (particularly e.g, acne, rosacea, eczema).
8. Subjects with history of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, medication, cosmetic or personal care products or ingredients.
9. Subject presenting a stable or progressive serious disease (per investigator's assessment).
10. Immuno-compromised subject.
11. Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).
12. Subjects regularly practicing aquatic or nautical sports.
13. Subjects regularly attending a sauna.
14. Subject with cardiovascular or circulatory history.
15. Subject with a history of skin cancer or malignant melanoma.
16. Intake of antihistamines, antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune-suppressants in the last 6 months before study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Clinical scoring for skin redness | Baseline, Time point post-induction 5 min , Time point post-intervention 5 min，Time point post-intervention 1 hour, Time point post-intervention 2 hours.
  Participants: N= 30
Clinical scoring for skin redness | Baseline, Time point post-induction 5 min.
  Participants: N= 30
Image Capture and Analysis（Redness area ratio） | Baseline, Time point post-induction 5 min , Time point post-intervention 5 min，Time point post-intervention 1 hour, Time point post-intervention 2 hours.
  Participants: N= 30，by VISIA 7
Image Capture and Analysis（Redness area ratio） | Baseline, Time point post-induction 5 min , Time point post-intervention 5 min，Time point post-intervention 1 hour, Time point post-intervention 2 hours.
  Participants: N= 30,by TiVi 700 Tissue Viability Imager
Instrumental Assessment (Erythema index) | Baseline, Time point post-induction 5 min , Time point post-intervention 5 min，Time point post-intervention 1 hour, Time point post-intervention 2 hours.
  Participants: N= 30, by Mexameter
Consumer Questionnaire | Time point post-intervention 10 sec, Time point post-intervention 1 min, Time point post-intervention 5 min，Time point post-intervention 1 hour, Time point post-intervention 2 hours.
  Participants: N= 60

CONTACTS AND LOCATIONS:
Overall Officials: Ping Xu, Principal Investigator — Shanghai China-norm Quality Technical Service Co., Ltd.
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
This Data Sharing Plan (DSP) aims to promote the open exchange and reuse of de-identified individual participant data (IPD) from cosmetic clinical research, including study protocols, case report forms (CRFs), and statistical analysis plans (SAPs). The shared data will be made available through compliant platforms to eligible researchers in dermatology, cosmetic science, and related fields, following ethical principles and data protection regulations. Users must sign a Data Use Agreement (DUA) to ensure data security, privacy protection, and compliance with research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18-Month Duration: The data sharing period starts upon study completion and PRS registration completion.
  Timeline:
  Months 2-3: Data de-identification, metadata preparation, and platform integration.
  Month 4: Official launch of data access.
Access Criteria: Primary Platform:
  ResMan (www.medresman.org.cn) - China's leading medical research data repository.
  Eligibility:
  Researchers/affiliates from academic institutions, hospitals, or registered research organizations.
  Engaged in dermatology, cosmetic science, or related fields. Able to demonstrate ethical compliance and data security capabilities.
URL: http://www.medresman.org.cn